CLINICAL TRIAL: NCT00215878
Title: D-serine for Posttraumatic Stress Disorder Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herzog Hospital (Other)
Responsible Party: Principal Investigator, Heresco-Levi Uriel, Principal Investigator, Herzog Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Heresco2CTIL; 20030311
Record Dates: First submitted 2005-09-18; First posted 2005-09-22 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Adjuvant 6 weeks treatment with placebo (~2g /day)
  Interventions: Drug: D-serine (~2g /day)
- 2 (Experimental): Adjuvant 6 weeks treatment with D-serine (~2g /day)
  Interventions: Drug: D-serine (~2g /day)

INTERVENTIONS:
Drug: D-serine (~2g /day) — Two 6 weeks treatment arms under a cross over design. In one arm adjuvant treatment with experimental medication (D-serine ~2g /day), in the second arm adjuvant treatment with placebo (~2g /day)

SUMMARY:
The aim of this study is to asses the effects of the NMDA receptor full agonist D-serine while used as adjuvant treatment for individuals suffering from chronic posttraumatic stress disorder (PTSD). Dysfunction of neurotransmission mediated at NMDA receptor plays a cardinal role in the pathophysiology of PTSD and PTSD patients typically suffer from cognitive dysfunctions and avoidance& depressive symptomatology that may be mediated by NMDA receptor function deficits.

Thus, enhancement of NMDA activity by using D-serine may be beneficial in the treatment of PTSD. The study design involves two 6 week periods during which the participants will be randomly assigned to receive treatment with D-serine (~2g /dy)and placebo. This design allows each participant the opportunity to respond to the experimental treatment.

ELIGIBILITY:
Inclusion Criteria:

• Chronic PTSD (DSM-IV diagnosis)

Exclusion Criteria:

* Other psychiatric diagnosis
* Substance abuse
* Unstable medical condition

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
CAPS scores | 6 week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Uriel Heresco-Levy, M.D, Principal Investigator — Ezrat Nashim-Herzog Memorial Hospital
Locations (1):
- Ezrat Nashim-Herzog Memorial Hospital, Jerusalem, Israel

REFERENCES:
- [Derived] Heresco-Levy U, Vass A, Bloch B, Wolosker H, Dumin E, Balan L, Deutsch L, Kremer I. Pilot controlled trial of D-serine for the treatment of post-traumatic stress disorder. Int J Neuropsychopharmacol. 2009 Oct;12(9):1275-82. doi: 10.1017/S1461145709000339. Epub 2009 Apr 15. PMID 19366490